CLINICAL TRIAL: NCT02912832
Title: TBDx Feasibility Study: Prospective Study to Determine the Feasibility of Automated Smear Microscopy
Brief Title: Prospective Assessment of TBDx Feasibility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 7012-05-3/1
Record Dates: First submitted 2016-09-09; First posted 2016-09-23 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Pulmonary Tuberculosis
Keywords: Diagnosis
MeSH Terms: conditions — Tuberculosis, Pulmonary; Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- TBDx (Experimental): All samples were tested with TBDx and compared with smear microscopy and Xpert MTB/RIF using solid and liquid culture as gold standard.
  Operators were blinded to all other results for a sample upon data entry.
  Interventions: Device: TBDx

INTERVENTIONS:
Device: TBDx — The TBDx is an automated platform is based on an Olympus BX41 microscope with a 40 x objective lens, fitted with an Olympus XC 10 colour camera and a movable slide stage, with an attached computer that receives high-quality digital images acquired from the camera. The computer then operates detection algorithms that segment, evaluate, and classify objects of interest in these images which can be stored for subsequent review. The platform is able to integrate an optional 200-slide automated slide loader for high volume settings. The application can capture 100, 300 or more digital fields-of-view and can provide results for positive or negative smears in 5 minutes or less.
  Other Names: Automated microscopy

SUMMARY:
The purpose of this study will be to determine the performance characteristics of TBDx with culture as a gold standard. In addition, the investigators will assess the laboratory technicians' appraisal and technical suitability of the TBDx system.

DETAILED DESCRIPTION:
This will be a blinded, prospective study to determine the performance of the TBDx system for detection of pulmonary TB in comparison to LED microscopy and culture as a gold standard. The study will involve recruitment of 300 TB suspects per site with a high workload and experienced technicians. Participants will be recruited under the FIND TB Reference Materials project and leftover sputum samples used for the assessment of the TBDx.

ELIGIBILITY:
Inclusion Criteria:

* Persistent cough (>2 weeks) and at least one other typical symptom of pulmonary TB (fever, night sweats, malaise, recent weight loss, contact with active case, hemoptysis, chest pain, loss of appetite)
* Provision of informed consent (FIND TB Reference Materials)
* Provision of sputum for adequate testing

Exclusion Criteria:

* Patients receiving any anti-TB medication, in the 60 days prior to testing.
* Patients with only extra-pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2014-10; Primary Completion 2015-03 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Performance of TBDx compared to culture | 6 months
  Sensitivity, specificity and predictive values of TBDx compared to two solid (Löwenstein Jensen) and two liquid (MGIT) cultures

SECONDARY OUTCOMES:
Training needs through questionnaire assessment | 6 months
  Two days of hands-on, onsite TBDx training was provided to laboratory technicians with prior experience using smear microscopy, followed by 1-day observation. Each operator performed 3-4 runs under supervision and a proficiency assessment was conducted prior to study initiation. Following study completion all technicians were given a survey to assess perception of training needs and ease of use.
Comparison of performance of TBDx on direct vs concentrated smear | 6 months
Performance of TBDx in combination with Xpert MTB/RIF through analysis of two different algorithms | 6 months
  The performance of an algorithm combining direct TBDx as a triage test, followed by Xpert for confirmation of positive TBDx cases for the different cut-off points was assessed
User appraisal regarding ease of use, hands-on-time and perceived benefit through appraisal questionnaire | 6 months
Identify potential difficulties for implementation through observation and user appraisal | 6 months
  Potential barriers for implementation were assessed through observation and appraisal questionnaires following study completion, taking into account total time, complexity, number of steps, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M Denkinger, MD, Study Director — Find
Locations (2):
- Instituto de Medicina Tropical Alexander von Humboldt - Universidad Peruana Cayetano Heredia, Lima, Peru
- Pham Ngoc Thach Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient and results dataset will be made available upon publication of study findings

REFERENCES:
- See also: TBDx Proof of concept — http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0050173